CLINICAL TRIAL: NCT02842164
Title: Foley's Catheter Balloon for Induction of Mid Trimester Abortion in Nulliparous Women With or Without Tension Applied
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIOA
Record Dates: First submitted 2016-07-15; First posted 2016-07-22 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Induction of Abortion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Foley Catheter Balloon with Tension group (Other): a 16 French transcervical Foley catheter balloon will be advanced to or past the internal os and the balloon will be filled. Then catheter will be placed on gentle traction by taping the distal tip to the medial thigh for maximum 24 hours. To maintain gentle traction, periodic repositioning of the distal tip on the thigh will be necessary.
  Interventions: Other: Tension group; Other: Foley catheter Balloon
- Foley Catheter Balloon without tension group (Other): The Foley catheter balloon will be just supported by simple taping to the thigh.
  Interventions: Other: No tension group; Other: Foley catheter Balloon

INTERVENTIONS:
Other: Tension group
  Arms: Foley Catheter Balloon with Tension group
Other: No tension group
  Arms: Foley Catheter Balloon without tension group
Other: Foley catheter Balloon

SUMMARY:
Induction of abortion is a hot subject that has complex and emotional controversy. The most common time of abortion is the second trimester which represent about 10-15% of all induced abortions over the world. As well as, two-thirds of all serious abortion-related complications are related to induced second trimester abortion.

There are many causes for induction of abortion in the second trimester such as missed abortion, serious fetal abnormalities such as central nervous system or skeletal malformation and lastly some women do not wish to continue a pregnancy and will often seek out termination of pregnancy.

Termination of second trimester is more risky than the first trimester. So many lines have been emerged to achieve safe and effective method of termination of second trimester.

Pharmacologic management seems to be an appealing method for induction of abortion. The combing between mifepristone and misoprostol is the effective regimen for termination of second trimester abortion with success rate reaching about 97-99% within 24 hours.

However, mifepristone is not available or affordable in many countries worldwide so misoprostol have been used alone but it needs higher total dose with lower effectiveness and higher percentage of side effects rate than the combined regimens.

The optimal method for inducing second trimester nulliparous women with an unfavorable cervix is not known. Several studies in literature have described the effectiveness of Foley's catheter in cervical ripening and improvement of Bishop's score in women with unripe cervices . It may act in addition to its mechanical effect by increasing the release of prostaglandin and/or oxytocin release secondary to localized inflammation.

In practice, the insertion of intra-cervical Foley's catheter balloon is followed by applying tension in trial to shorten the time between the insertion and expulsion of the fetus, however; this tension adds more pain for the pregnant women with higher rate of vaginal bleeding and dissatisfaction.

Gary et al in 2016 concluded that the application of tension did not result in faster delivery times, but did result in faster times to catheter expulsion.

ELIGIBILITY:
Inclusion Criteria:

* Singleton second trimester (12-28 weeks) pregnancy.
* Nulliparous woman.
* Bishop score ≤ 6.
* BMI 18-22.5 kg/m2

Exclusion Criteria:

* Multiple gestations.
* Premature rupture of membranes before induction.
* Pregnancy complicated by antepartum hemorrhage (placenta previa or abruptio placenta).
* Low amniotic fluid volume (< 5cm).
* Scarred uterus including hysterotomy or myomectomy.
* Uterine infection.
* Unexplained bleeding.
* Latex allergy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The degree of pain provoked by catheter measured by visual analogue scale | 6 hours

SECONDARY OUTCOMES:
The time from insertion of Foley catheter balloon to catheter expulsion. | 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes